CLINICAL TRIAL: NCT07374250
Title: Perioperative Ivonescimab Plus S-1 and Oxaliplatin (SOX) Versus SOX Alone for Locally Advanced Gastric or GEJ Adenocarcinoma: A Multicenter Randomized Phase II Study
Brief Title: Perioperative Ivonescimab Plus S-1 and Oxaliplatin (SOX) for Locally Advanced Gastric or GEJ Adenocarcinoma
Acronym: Huaxi
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Bo Zhang, MD, Chief Physician, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Huaxi gastric cancer; Huaxi (Other: Huaxi)
Record Dates: First submitted 2025-12-10; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; RCT
Keywords: gastric cancer; Ivonescimab; neoadjuvant treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Ivonescimab Plus S-1 and Oxaliplatin (SOX)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOX (Active Comparator): oxaliplatin, S-1, four 3-week cycles were administered.
  Interventions: Drug: Oxaliplatin; Drug: S-1
- ISOX (Experimental): In the ISOX group, the regimen included ivonescimab, oxaliplatin, and S-1.
  Interventions: Drug: Ivonescimab (20mg/kg Q3W); Drug: Oxaliplatin; Drug: S-1

INTERVENTIONS:
Drug: Ivonescimab (20mg/kg Q3W) — ivonescimab (20 mg/kg), four 3-week cycles were administered; ivonescimab was not administered in cycle 4. .
  Arms: ISOX
Drug: Oxaliplatin — Oxaliplatin (130 mg/m², administered intravenously on day 1), four 3-week cycles were administered.
Drug: S-1 — S-1 (administered orally twice daily on days 1-14 of each 21-day cycle, with the daily dose determined by body surface area: <1.25 m², 80 mg/day; ≥1.25 to <1.5 m², 100 mg/day; ≥1.5 m², 120 mg/day), four 3-week cycles were administered.

SUMMARY:
The purpose of this clinical trial is to evaluate whether perioperative ivonescimab in combination with S-1 and oxaliplatin (SOX) is effective in treating locally advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma. The study will also assess the safety profile of this treatment regimen.

Primary Objective:

To determine whether perioperative ivonescimab plus SOX improves the pathological complete response (pCR) rate compared with SOX alone in patients with locally advanced gastric or GEJ adenocarcinoma.

Study Design:

Participants will be randomly assigned to receive either ivonescimab plus SOX or SOX alone to evaluate the potential added benefit of ivonescimab in this setting.

Participation Details:

Participants will receive the assigned treatment (ivonescimab plus SOX or SOX alone) every 21 days for approximately 4 months.

They will visit the clinic once every 3 weeks for evaluations, laboratory tests, and monitoring.

Participants will be asked to keep a daily diary to record any symptoms or side effects experienced during the study.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of ivonescimab in combination with S-1 and oxaliplatin (SOX) for the treatment of locally advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma in the neoadjuvant (perioperative) setting, with the goal of improving the pathological complete response (pCR) rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Histologically confirmed gastric or gastroesophageal junction (G/GEJ) adenocarcinoma.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Clinically staged as T3-4a N+ M0 by computed tomography (CT) or magnetic resonance imaging (MRI).
5. Considered eligible for curative resection.
6. No prior antitumor therapy for the current disease.
7. Adequate organ function, including hepatic, renal, and bone marrow function, as per prespecified laboratory criteria.
8. Expected survival of ≥6 months.

Exclusion Criteria:

1. Known mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) tumor.
2. Uncontrolled hypertension, defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥ 90 mmHg despite optimized antihypertensive therapy, or hypertension complicated by acute events (e.g., hypertensive crisis, hypertensive encephalopathy) that cannot be stably controlled.
3. Tumor lesions with a bleeding tendency, including but not limited to: active ulcerative tumor lesions, hematemesis within 2 months prior to informed consent, high risk of major gastrointestinal bleeding as determined by the investigator.
4. History of thromboembolic or arterial/venous vascular events within 6 months prior to enrollment, such as cerebrovascular events (including transient ischemic attack), deep vein thrombosis, or pulmonary embolism.
5. Gastrointestinal perforation or gastrointestinal obstruction within 6 months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (pCR; ypT0) assessed by investigators, defined as the complete absence of tumor cells in the primary tumor on pathological examination. | Perioperative

SECONDARY OUTCOMES:
Event-free survival (EFS) | Through study completion,an average of 2 years
  Event-free survival (EFS), defined as the time from randomization to the first occurrence of relapse, metastasis, or death from any cause;
major pathologic response | Perioperative
  defined as ≤10% residual viable tumor cells in the resected primary tumor specimen after neoadjuvant therapy;
R0 resection | Perioperative
  defined as microscopically margin-negative resection
overall survival (OS) | Through study completion,an average of 2 years
  defined as the time from randomization to death from any cause;
disease-free survival (DFS) | Through study completion,an average of 2 years
  defined as the time from the post-surgery baseline scan to the first occurrence of relapse, metastasis, or death from any cause
safety | Through study completion,an average of 2 years
  Treatment-related adverse events (TRAEs) with potential immunologic etiology were categorized and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) (Version 5.0)
surgery-related complications | Through study completion,an average of 2 years
  were graded according to the Clavien-Dindo classification;
An exploratory endpoint | Through study completion,an average of 2 years
  was the evaluation of potential predictive biomarkers associated with treatment response
Quality of life | Perioperative
  Quality of life was assessed using the EORTC QLQ-STO22 and EORTC QLQ-C30 questionnaires, administered at three time points: within one week before initiation of neoadjuvant therapy, within one week before the fourth neoadjuvant therapy cycle, and at 30 days postoperatively (±3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Gou Hongfeng, Principal Investigator — Gastric Cancer Center, West China Hospital, Sichuan University, 37 Guoxue Alley, Chengdu 610041, Sichuan, China.
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) may not be shared due to privacy and confidentiality concerns, legal or ethical restrictions, limitations in data sharing agreements or consent, intellectual property rights, commercial interests, or because of technical and resource constraints related to data anonymization and sharing.

REFERENCES:
- [Result] Andre T, Tougeron D, Piessen G, de la Fouchardiere C, Louvet C, Adenis A, Jary M, Tournigand C, Aparicio T, Desrame J, Lievre A, Garcia-Larnicol ML, Pudlarz T, Cohen R, Memmi S, Vernerey D, Henriques J, Lefevre JH, Svrcek M. Neoadjuvant Nivolumab Plus Ipilimumab and Adjuvant Nivolumab in Localized Deficient Mismatch Repair/Microsatellite Instability-High Gastric or Esophagogastric Junction Adenocarcinoma: The GERCOR NEONIPIGA Phase II Study. J Clin Oncol. 2023 Jan 10;41(2):255-265. doi: 10.1200/JCO.22.00686. Epub 2022 Aug 15. PMID 35969830
- [Result] Lorenzen S, Gotze TO, Thuss-Patience P, Biebl M, Homann N, Schenk M, Lindig U, Heuer V, Kretzschmar A, Goekkurt E, Haag GM, Riera-Knorrenschild J, Bolling C, Hofheinz RD, Zhan T, Angermeier S, Ettrich TJ, Siebenhuener AR, Elshafei M, Bechstein WO, Gaiser T, Loose M, Sookthai D, Kopp C, Pauligk C, Al-Batran SE; AIO and SAKK Study Working Groups. Perioperative Atezolizumab Plus Fluorouracil, Leucovorin, Oxaliplatin, and Docetaxel for Resectable Esophagogastric Cancer: Interim Results From the Randomized, Multicenter, Phase II/III DANTE/IKF-s633 Trial. J Clin Oncol. 2024 Feb 1;42(4):410-420. doi: 10.1200/JCO.23.00975. Epub 2023 Nov 14. PMID 37963317
- [Result] Shah MA, Kennedy EB, Alarcon-Rozas AE, Alcindor T, Bartley AN, Malowany AB, Bhadkamkar NA, Deighton DC, Janjigian Y, Karippot A, Khan U, King DA, Klute K, Lacy J, Lee JJ, Mehta R, Mukherjee S, Nagarajan A, Park H, Saeed A, Semrad TJ, Shitara K, Smyth E, Uboha NV, Vincelli M, Wainberg Z, Rajdev L. Immunotherapy and Targeted Therapy for Advanced Gastroesophageal Cancer: ASCO Guideline. J Clin Oncol. 2023 Mar 1;41(7):1470-1491. doi: 10.1200/JCO.22.02331. Epub 2023 Jan 5. PMID 36603169
- [Result] Chao J, Fuchs CS, Shitara K, Tabernero J, Muro K, Van Cutsem E, Bang YJ, De Vita F, Landers G, Yen CJ, Chau I, Elme A, Lee J, Ozguroglu M, Catenacci D, Yoon HH, Chen E, Adelberg D, Shih CS, Shah S, Bhagia P, Wainberg ZA. Assessment of Pembrolizumab Therapy for the Treatment of Microsatellite Instability-High Gastric or Gastroesophageal Junction Cancer Among Patients in the KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Clinical Trials. JAMA Oncol. 2021 Jun 1;7(6):895-902. doi: 10.1001/jamaoncol.2021.0275. PMID 33792646
- [Result] Nie RC, Chen GM, Yuan SQ, Kim JW, Zhou J, Nie M, Feng CY, Chen YB, Chen S, Zhou ZW, Wang Y, Li YF. Adjuvant Chemotherapy for Gastric Cancer Patients with Mismatch Repair Deficiency or Microsatellite Instability: Systematic Review and Meta-Analysis. Ann Surg Oncol. 2022 Apr;29(4):2324-2331. doi: 10.1245/s10434-021-11050-6. Epub 2021 Nov 18. PMID 34796431
- [Result] Choi YY, Bae JM, An JY, Kwon IG, Cho I, Shin HB, Eiji T, Aburahmah M, Kim HI, Cheong JH, Hyung WJ, Noh SH. Is microsatellite instability a prognostic marker in gastric cancer? A systematic review with meta-analysis. J Surg Oncol. 2014 Aug;110(2):129-35. doi: 10.1002/jso.23618. Epub 2014 Apr 15. PMID 24737677
- [Result] Pietrantonio F, Miceli R, Raimondi A, Kim YW, Kang WK, Langley RE, Choi YY, Kim KM, Nankivell MG, Morano F, Wotherspoon A, Valeri N, Kook MC, An JY, Grabsch HI, Fuca G, Noh SH, Sohn TS, Kim S, Di Bartolomeo M, Cunningham D, Lee J, Cheong JH, Smyth EC. Individual Patient Data Meta-Analysis of the Value of Microsatellite Instability As a Biomarker in Gastric Cancer. J Clin Oncol. 2019 Dec 10;37(35):3392-3400. doi: 10.1200/JCO.19.01124. Epub 2019 Sep 12. PMID 31513484
- [Result] Tran-Minh ML, Lehmann-Che J, Lambert J, Theou-Anton N, Pote N, Dior M, Mary F, Goujon G, Gardair C, Schischmanoff O, Kaci R, Cucherousset N, Bertheau P, Couvelard A, Aparicio T; for NORDICAP. Prevalence and prognosis of microsatellite instability in oesogastric adenocarcinoma, NORDICAP 16-01. Clin Res Hepatol Gastroenterol. 2021 Jul;45(4):101691. doi: 10.1016/j.clinre.2021.101691. Epub 2021 Apr 20. PMID 33852952
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Arnold M, Ferlay J, van Berge Henegouwen MI, Soerjomataram I. Global burden of oesophageal and gastric cancer by histology and subsite in 2018. Gut. 2020 Sep;69(9):1564-1571. doi: 10.1136/gutjnl-2020-321600. Epub 2020 Jun 30. PMID 32606208